CLINICAL TRIAL: NCT01792492
Title: The Role of an Optical Probe in the Detection of Thyroid Cancer and Normal Thyroid Tissue in a Thyroidectomy Specimen: A Pilot Study
Brief Title: The Role of an Optical Probe in Thyroid Cancer Diagnosis: Pilot Study
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Stephanie Lee, Assistant Professor of Medicine, Boston Medical Center
Other Study IDs: H28135
Record Dates: First submitted 2011-07-08; First posted 2013-02-15 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Thyroid Nodule; Thyroid Neoplasms; Thyroid Cancer
Keywords: Thyroid Neoplasms; Optical Devices; Spectrum Analysis; Thyroid diseases
MeSH Terms: conditions — Thyroid Nodule; Thyroid Neoplasms; Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will investigate the usefulness of an optical probe in the differentiation of thyroid cancer from normal thyroid tissue in a thyroidectomy specimen.

DETAILED DESCRIPTION:
The optical real-time readings will be compared to the histological analysis from the same area. Subjects undergoing thyroid surgery for thyroid disease including thyroid nodules, thyroid cancer and thyroid goiter with nodules will be eligible to participate. After the removal of the thyroid gland, optical readings will be taken from the ex vivo thyroid gland and these same areas will then be analyzed in the usual standard fashion. The reading will then be correlated with the histological results. In addition, if lymph nodes are removed as part of the surgery they will also be tested prior to histological standard processing. All specimens and data will be de-identified.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing thyroid surgery for thyroid nodules, thyroid cancer, and thyroid goiter with nodules.

Exclusion Criteria:

* Subjects whose thyroid specimens have been put in formalin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Tertiary hospital setting Urban hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-06; Primary Completion 2010-03 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Assess optical probe for the differentiation of thyroid cancer from normal thyroid tissue and benign thyroid nodules | two years
  The objective is to assess a device called an optical probe for the differentiation of thyroid cancer from normal thyroid tissue, benign thyroid nodules or parathyroid glands, and the detection of thyroid cancer within lymph nodes using a hand-held spectroscope, compare the spectra from benign and malignant thyroid nodules and use this to discriminate benign from malignant nodules based on final histopathology or cytology as the gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Rosen, M.D. FACS, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No